CLINICAL TRIAL: NCT05143112
Title: Allogeneic CD19 CAR-T Cells for the Treatment of Relapsed/Refractory B-cell Lymphoma
Acronym: CAR-T
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Professor, Shenzhen University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ONCO-008
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-02

CONDITIONS: Non-hodgkin Lymphoma,B Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Allogeneic CD19 CR-T cell infusion
  Interventions: Biological: Allogeneic CD19 CR-T cell

INTERVENTIONS:
Biological: Allogeneic CD19 CR-T cell — Allogeneic CD19 CR-T cell infusion

SUMMARY:
Preclinical and clinical studies of CD19 CAR-T in r/r B-NHL have been extensively carried out. At the beginning of 2020, MorphoSys submitted its company-targeted CD19 monoclonal antibody to the FDA for r/r DLBL treatment and obtained FDA priority approval. It further confirms the safety and effectiveness of CD19 as a therapeutic target in r/r B-NHL. However, these CAR-T cells are constructed from patients' autologous T cells, and the production and preparation time is long; on the other hand, most patients have received multiple chemotherapy before CAR-T treatment, and the quantity and quality of T cells often cannot meet the needs of clinical treatment. It is also an important factor leading to the failure of CAR-T cell therapy, which limits the large-scale clinical application of CAR-T.

T cells sourced from healthy people are not only sufficient in quantity and quality guaranteed, but also available at any time. In December 2020, lancet[2] reported a clinical study of 19 patients receiving allogeneic CAR-T cell therapy for B-ALL. 14 patients were evaluated as CR/CRi (67%) 28 days after treatment, with a median sustained remission Time 4.1 months. Allogeneic CAR-T cells are safe and effective for the treatment of B-cell malignant diseases, and their clinical application range is expected to further improve the remission rate and survival rate of patients with R/R B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR) T cells enable T cells to recognize and kill tumor cells that express specific antigens through genetic engineering. CD19 is expressed on the membrane surface of pre-B cells and mature B cells, but not on the surface of T cells and normal granulocytes. It is an ideal therapeutic target for B cell-derived tumors. A large number of previous studies have confirmed that CD19 CAR-T cells are a safe and effective method for the treatment of ALL. In 2019, Locke FL[1] et al. reported a clinical study of CD19 CAR-T for r/r DLBL. 119 patients were enrolled. The objective response rate was 83%, the CR rate was 58%, and the median progression-free survival was 5.9. Months. Greatly improved the patient's prognosis.

Preclinical and clinical studies of CD19 CAR-T in r/r B-NHL have been extensively carried out. At the beginning of 2020, MorphoSys submitted its company-targeted CD19 monoclonal antibody to the FDA for r/r DLBL treatment and obtained FDA priority approval. It further confirms the safety and effectiveness of CD19 as a therapeutic target in r/r B-NHL. However, these CAR-T cells are constructed from patients' autologous T cells, and the production and preparation time is long; on the other hand, most patients have received multiple chemotherapy before CAR-T treatment, and the quantity and quality of T cells often cannot meet the needs of clinical treatment. It is also an important factor leading to the failure of CAR-T cell therapy, which limits the large-scale clinical application of CAR-T.

T cells sourced from healthy people are not only sufficient in quantity and quality guaranteed, but also available at any time. In December 2020, lancet[2] reported a clinical study of 19 patients receiving allogeneic CAR-T cell therapy for B-ALL. 14 patients were evaluated as CR/CRi (67%) 28 days after treatment, with a median sustained remission Time 4.1 months. Allogeneic CAR-T cells are safe and effective for the treatment of B-cell malignant diseases, and their clinical application range is expected to further improve the remission rate and survival rate of patients with R/R B-cell non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. 14-70 years old (including 14, 70 years old), no gender limit;
2. According to the 2020 World Health Organization (WHO) diagnostic criteria, it is diagnosed as relapsed/refractory B-cell non-Hodgkin lymphoma (R/R B-NHL);
3. The ECOG behavior status score is 0-2 points;
4. Expected survival time ≥ 3 months;
5. Tumor cells express CD19;
6. Those who have failed autologous CAR-T cell preparation or autologous CAR-T cell therapy under the existing technical conditions;
7. No serious heart, lung, liver, or kidney disease;
8. Ability to understand and willing to sign the informed consent form for this trial.

Cell donors must meet the following criteria to participate in this study:

1. 18-60 years old, no gender limit;
2. A fully matched/half-matched donor with the patient's HLA match;

9) No contraindications to peripheral blood apheresis

Exclusion Criteria:

1. Tumor cells do not express CD19;
2. Active infection;
3. Abnormal liver function (total bilirubin>1.5×ULN, ALT>2.5×ULN), abnormal renal function (serum creatinine>1.5×ULN);
4. People with unstable angina or New York Heart Association class 3/4 congestive heart failure, multiple organ dysfunction;
5. HIV/AIDS patients;
6. Those who need long-term anticoagulation (warfarin or heparin), antiplatelet (aspirin, dose>300mg/d; clopidogrel, dose>75mg/d) treatment;
7. Those who received radiotherapy within 4 weeks before the start of the study (blood sampling);
8. Known or suspected drug abuse or alcohol dependence;
9. People with mental illness or other conditions cannot obtain informed consent, and cannot cooperate with the requirements of completing the experimental treatment and inspection procedures;
10. Participated in other clinical trials within 30 days;
11. Pregnant or lactating women, male subjects (or their partners) or female subjects have a pregnancy plan during the study period to 6 months after the end of the test, and are unwilling to use a medically approved effective contraceptive measure during the test period (Such as intrauterine contraceptive devices or condoms);
12. Those who are judged by the investigator to be unsuitable to participate in this trial

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | From date of initial treatment to the end of follow up, up to 2 years
  Percentage of patients in complete remission in total treated patients

SECONDARY OUTCOMES:
overall survival rate | From admission to the end of follow up, up to 2 years
  Time from initiation of trial treatment to death

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Dr, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Li Yu, Shenzhen, Guangdong, China